CLINICAL TRIAL: NCT05203835
Title: A Pilot Placebo-Controlled Trial of Acebilustat (CTX-4430) for the Treatment of Human Upper Extremity Lymphedema
Brief Title: Trial of Acebilustat for the Treatment of Upper Arm Lymphedema
Acronym: HEAL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Celltaxis LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-62051; NCI-2022-09343 (Other: CTRP); BRS0140 (Other: OnCore)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lymphedema of Upper Arm
MeSH Terms: interventions — acebilustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Placebo and acebilustat (Experimental): Participants will take acebilustat and placebo over a period of 9 months.
  Interventions: Drug: Acebilustat; Drug: Placebo

INTERVENTIONS:
Drug: Acebilustat — By mouth, once a day, 100 mg capsule
Drug: Placebo — Placebo to match acebilustat by mouth, once a day

SUMMARY:
This study is designed to investigate the response of unilateral upper extremity (arm) lymphedema, during pharmacologic treatment of lymphedema with oral placebo and oral acebilustat. Participants will receive "study drug" (Acebilustat or placebo), for 9 months. For 3 of these months, the participant will receive placebo; for 6 of these months, the participant will receive active ingredient, acebilustat. The study is blinded which means that the participant will not be told which study pill they are taking.

DETAILED DESCRIPTION:
To enter this study, participants will have to meet requirements that will be evaluated during screening, Visit 1. If eligible, and if they choose to continue, Visit 2, treatment start, will take place 2-7 days later. Study visits are every (approximately) 90 days. Physical exam, including limb measurements and skin measurements (with tape measure and dermal ultrasound) are performed. Phlebotomy for research samples and clinical labs will be performed at study start and end of study.

ELIGIBILITY:
Inclusion Criteria:

* Upper arm lymphedema, single arm, stage 2, greater than 6 months duration
* Male or female.
* Ages 18-75.
* Prior imaging by lymphoscintigraphy or magnetic resonance lymphangiography that confirms the presence of lymphedema in the affected limb OR, at screening, an affected:unaffected limb volume ratio of ≥1.1 with significant history of lymphedema
* Consistent use of an appropriately sized compression garment for daytime use.
* Willing to maintain a stable regimen of self-care from screening to end-of-study.
* If a potential participant has undergone prior microvascular (vascular lymph node transfer, lymphaticovenous anastomosis) or debulking surgical intervention, at least one year must have elapsed prior to screening AND, at screening, an affected: unaffected limb volume ratio of ≥1.1.
* Lymphedema therapy must be completed at least 8 weeks prior to screening.
* Has received Covid-19 vaccine (Pfizer, Moderna or Johnson & Johnson)
* Ability to understand and the willingness to sign a written informed consent document.
* . If the possibility of conception exits, agrees to use a medically acceptable method of contraception (both male and female) from the signing of the informed consent form through the entire study period; men or women who are surgically sterile (> 6 months after surgery) or women who have been postmenopausal for at least 1 year are not considered to be of childbearing potential.

Exclusion Criteria:

* Concurrent participation in a clinical trial of any other investigational drug or therapy
* Other medical condition that could lead to acute limb edema (e.g. acute blood clot) or other medical condition that could result in symptoms overlapping those of lymphedema (e.g. frozen shoulder).
* History of clotting disorder.
* Chronic (persistent) infection in the affected limb.
* Active cancer treatment or history of cancer treatment within the past 2 years, except for non-melanoma skin cancer or cervical cancer in-situ.
* Chronic kidney disease
* Liver disease
* Pregnancy or nursing.
* Substance abuse (e.g., alcohol or drug abuse) within 6 months prior to screening.
* Any current use of non-steroidal anti-inflammatory drug (NSAID), e.g. ibuprofen, ketoprofen) or prior therapeutic use of ketoprofen.
* Any current use of immunosuppressive or immunomodulatory drugs (e.g., immunosuppressants, anticancer drugs, interleukins, interleukin antagonists or interleukin receptor blockers) or leukotriene pathway inhibitor (zileuton), leukotriene receptor antagonist (e.g montelukast).
* Personal or family history of prolonged QT syndrome
* Any reason (in addition to those listed above) that, in the opinion of the investigator, precludes full participation in the study.
* Any current use of statin drugs. The use of any statin drug should be discontinued at least 2 weeks prior to the trial enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in cutaneous thickness in the affected upper extremity, as measured by skin calipers. | Comparison of the measurement of week 0 to week 12 and of week 12 to week 36
  Cutaneous thickness will be measured by skin calipers at three designated locations in the affected upper extremity.

SECONDARY OUTCOMES:
Change in cutaneous dimensions and architecture in the affected upper extremity, as measured by ultrasound | Comparison of the measurement of week 0 to week 12 and of week 12 to week 36
  Cutaneous measurements will be derived from serial ultrasonographic examination at three designated locations in the affected upper extremity using a Terason 3200T device
Change in the volume of the affected upper extremity. | Comparison of the measurement of week 0 to week 12 and of week 12 to week 36.
  Volume changes in the affected upper extremity will be calculated through circumferential measurements of the limb and quantitated with the truncated cone approximation.
Change in LymQoL score | Comparison of the measurement of week 0 to week 12 and of week 12 to week 36.
  Change in the LymQoL (Lymphedema Quality of Life) questionnaire score will be used to assess the impact of lymphedema on patients' quality of life. The LymQoL is a validated, disease-specific tool measuring physical, psychological, appearance, and functional domains (range 0-100; higher scores indicate worse QoL).
Change in LymVAS score | Comparison of the measurement of week 0 to week 12 and of week 12 to week 36.
  Change in the LymVAS (Lymphedema Visual Analog Scale) questionnaire score will be used to assess patient-perceived lymphedema severity (0 = none, 10 = worst).

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Rockson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No